Study Title: Body Fat Reducing Effect and Safety of Enzymatically Modified Isoquercitrin in Obses

Subjects

PI: Mohsen Meydani Statistical Analysis Plan Version Date 3/2/2018

**Version Date:** 3/2/2018

Principal Investigator: Mohsen Meydani

**Co-Investigator:** Susan Roberts

Study Physician: Lisa Ceglia

Study Title: Body Fat Reducing Effect and Safety of Enzymatically Modified Isoquercitrin in Obese

Subjects

NCT Number: NCT02818699

## **Statistical Analysis Plan**

All subjects who completed the study were included in the analysis. Summary statistics were expressed in mean  $\pm$  S.D. for continuous variables, and counts (percentage %) for categorical variables. Differences between treatment groups were tested using Student's t-test. Two-sample Wilcoxon test is used when variables appear to violate distributional assumptions. Model assumptions were assessed within an ANCOVA model predicting 12 week outcome, adjusting for baseline. Fisher's exact test or chi-square test was performed for categorical variables. An  $\alpha$  level of p<0.05 was considered statistically significant. Statistical analysis was conducted in R 3.4 (R Core Team 2017, Vienna Austria).